CLINICAL TRIAL: NCT05279781
Title: Quality of Life, Satisfaction and Outcome After Full Pulpotomy Compared to Root Canal Therapy
Brief Title: Outcome of Pulpotomy Versus Root Canal Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 375/2019
Record Dates: First submitted 2021-11-23; First posted 2022-03-15 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Caries; Pulpitis - Irreversible
MeSH Terms: interventions — Pulpotomy

STUDY DESIGN:
Intervention Model Description: Two groups. One will receive root canal treatment t and the other will receive pulpotomy.
Who Masked: Participant
Masking Description: Participant will not be informed whether complete pulp removal or partial treatment was done.
  Operator and investigator cannot be blinded due to differences in the procedure and it will be evident on the radiographs, so it cannot be masked during radiographic evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Root canal treatment group (Active Comparator): This group will receive complete root canal therapy
  Interventions: Procedure: Non surgical root canal treatment
- Pulpotomy group (Active Comparator): This group will receive full pulpotomy
  Interventions: Procedure: Pulpotomy

INTERVENTIONS:
Procedure: Non surgical root canal treatment — Complete root canal treatment will be performed followed by direct restoration
  Arms: Root canal treatment group
Procedure: Pulpotomy — Full pulpotomy followed by direct restoration
  Arms: Pulpotomy group

SUMMARY:
Root canal therapy (RCT) is indicated once the pulp is diagnosed with irreversible pulpitis. Despite favorable success rate reported for RCT in vital cases, it is time consuming, and might increases fracture susceptibility of teeth. With the advancement of materials and better understanding of pulpal healing, vital pulp therapy is practiced as an alternative treatment with high success rate. The aim of this study is to explore the outcome, quality of life and patient satisfaction after full pulpotomy compared to RCT.

DETAILED DESCRIPTION:
Permanent molar teeth with carious pulp exposure and mature roots as evident on the preoperative periapical radiograph will be included in the study. The teeth will be randomly divided into 2 groups (n=30). The first group will be treated with Biodentine full pulpotomy and the second group will be endodontically treated. Based on a previously validated questionnaire. The quality of life and satisfaction of patients after pulpotomy treatment will be evaluated compared to those after endodontic treatment. Clinical and radiographic assessment of the treated teeth will be done 3, 6 and 12 months postoperatively. Pain level will be recorded preoperatively and 1, 2, 3, 5 and 7 days after treatment.

The questionnaire consists of five components:

1. Characteristics of the patient; including age, gender, socioeconomic status, smoking, oral hygiene practices, frequency of dental visits, and dental history.
2. Postoperative complications including postoperative pain, discomfort,or swelling.

   These symptoms will be evaluated after 1, 2, 3,5 and 7 days by contacting the patient on the phone and at follow up visits at 3, 6, and 12 months.
3. Quality of life instruments designed
4. Semantic scales designed to evaluate patient satisfaction with the treatment received.

Clinical and radiographic assessment of the treated teeth will be recorded. Success will be defined as clinically asymptomatic tooth with no sinus tract or swelling or periapical lesion.

Data will be analysed statistically using appropriate tests based on the distribution of the results.

ELIGIBILITY:
Inclusion Criteria:

* Medically fit patient
* mature permanent tooth with deep caries
* diagnosis of irreversible pulpits.
* tooth is restored with a direct restoration

Exclusion Criteria:

* immature teeth
* teeth were hemostasis cannot be achieved after pulpotomy
* necrotic teeth
* lack of response to cold test

Ages: 9 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-09-20 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Post operative pain level on numerical pain scale | 7 days
  Pain level after treatment will be assessed on a numerical scale from 0-10 where is zero refer to no pain and 10 is the most sever pain.
Post operative pain level on visual analogue scale | 7 days
  Pain level after treatment will be assessed on a visual analogy scale from 0-10, where is zero refer to no pain and 10 is the most sever pain.

SECONDARY OUTCOMES:
Clinical success | 6, 12, 24, 48 months
  The tooth should be pain free, no sinus tract, no tenderness to palpation and no swelling. As measured by clinical examination
Radiographic success | 6, 12, 24, 48 months
  Periapical x-ray will be taken it should show no bone lesions or root resorption

OTHER OUTCOMES:
The quality of life questionnaire | 6,12, 24, 48 months
  A questionnaire validated previously by Dugas et al 2002 will be used to assess Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Nessrin Taha, PhD, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan University of science and technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No
After collection of data and publication , data might be made available for the benefit off other researchers

REFERENCES:
- [Result] Taha NA, About I, Sedgley CM, Messer HH. Conservative Management of Mature Permanent Teeth with Carious Pulp Exposure. J Endod. 2020 Sep;46(9S):S33-S41. doi: 10.1016/j.joen.2020.06.025. PMID 32950193